CLINICAL TRIAL: NCT07027592
Title: The Relationship Between Training Dynamics and General Health Status With Injury Risk in Veteran Football Players
Brief Title: The Relationship Between Training Dynamics and General Health Status in Veteran Football Players
Status: Recruiting | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, AYŞE KAYALI VATANSEVER, Assistant Professor, Izmir Bakircay University
Other Study IDs: 25-4T/16
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Football; Injury; Veteran
Keywords: FIFA 11+; Veteran Football Players; Injury risk
MeSH Terms: conditions — Wounds and Injuries | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey Study — The injury risk in veteran football players will be assessed based on FIFA 11+.

SUMMARY:
The goal of this observational study is to learn how training habits and general health status are related to injury risk in veteran football players (men over 35 years old who play recreational football). The main questions it aims to answer are:

Do specific training patterns (such as frequency, intensity, and duration) increase or lower the risk of injury?

How does general health status (including factors like sleep, nutrition, and existing health conditions) affect injury risk?

Participants will:

Complete questionnaires about their training habits, lifestyle, and general health

Report any injuries they experience during the football season

Attend periodic health assessments

ELIGIBILITY:
Inclusion Criteria:

* Playing football as a veteran

Exclusion Criteria:

* Not participating in a regular training program

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veteran football players
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Injury Rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No